CLINICAL TRIAL: NCT03567005
Title: Clinical Validation of DACP Digital Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLD523-C001
Record Dates: First submitted 2018-06-13; First posted 2018-06-25 (Actual); Results first posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-05

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- DACP Digital then DACP (Other): Nelfilcon A digital contact lenses worn first, followed by nelfilcon A contact lenses. Each product worn bilaterally (in both eyes) for 7 days in a daily disposable modality.
  Interventions: Device: Nelfilcon A digital contact lenses; Device: Nelfilcon A contact lenses
- DACP then DACP Digital (Other): Nelfilcon A contact lenses worn first, followed by nelfilcon A digital contact lenses. Each product worn bilaterally for 7 days in a daily disposable modality.
  Interventions: Device: Nelfilcon A digital contact lenses; Device: Nelfilcon A contact lenses

INTERVENTIONS:
Device: Nelfilcon A digital contact lenses — Silicone hydrogel digital contact lenses
  Other Names: DAILIES® AquaComfort Plus® Digital; DACP Digital
Device: Nelfilcon A contact lenses — Silicone hydrogel spherical contact lenses
  Other Names: DAILIES® AquaComfort Plus®; DACP

SUMMARY:
The purpose of this study is to evaluate the visual performance of DAILIES® AquaComfort Plus® (DACP) Digital lenses by assessing distance visual acuity (VA) as compared to DACP sphere contact lenses after one week of wear.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign an IRB/IEC approved Informed Consent form;
* Current wearer of DACP spherical contact lenses (at least 2 months in current correction), with a minimum wearing time of 5 days per week and 8 hours per day;
* Experiencing symptoms of eye strain from using technology;
* Willing to wear study lenses each day;
* Possess spectacles that provide a corrected visual acuity of 20/40 or better in both eyes (OU) and be willing to wear them (as needed);
* Willing to NOT use rewetting/lubricating drops at any time during the study;
* Currently using digital devices (computer, tablet, and/or smart phone) for a minimum of 5 days per week and 4 hours per day;
* Willing to NOT use any near aid (e.g. reading glasses) at any time during the study.

Exclusion Criteria:

* Conditions, use of medications, injury, or surgery, as specified in the protocol;
* Wearing habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment;
* Monocular (only one eye with functional vision);
* Pregnant.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2018-08-26 (Actual); Study Completion 2018-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon Research, Study Director — Alcon Research
Locations (4):
- United States (4):
  - Alcon Investigative Site, Bloomington, Illinois
  - Alcon Investigative Site, Powell, Ohio
  - Alcon Investigative Site, Brentwood, Tennessee
  - Alcon Investigative Site, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 5 investigative sites located in the United States.
Pre-assignment Details: All 60 enrolled subjects were randomized and exposed to the investigational products.
Period: Period 1, First 7 Days of Wear
Arm/Group | DACP Digital Then DACP | DACP Then DACP Digital
Started | 29 | 31
Completed | 29 | 31
Not Completed | 0 | 0
Period: Period 2, Second 7 Days of Wear
Arm/Group | DACP Digital Then DACP | DACP Then DACP Digital
Started | 29 | 31
Completed | 29 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects who were exposed to any study lenses evaluated in this study (Full Analysis Set).
Groups:
- Overall: Nelfilcon A digital contact lenses and nelfilcon A contact lenses worn during Period 1 and Period 2 in a crossover assignment, as randomized.
Arm/Group | Overall
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.2 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 56
  Black or African American | 3
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Distance Visual Acuity (VA) (logMAR, OU)
Description: VA was tested under photopic (well-lit) conditions using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart positioned 6 meters from the subject. VA was collected bilaterally (OU) and measured in logMAR (logarithm of the minimum angle of resolution), with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on the ETDRS chart. A lower numeric value represents better visual acuity.
Time Frame: Day 7, each product
Population: Full Analysis Set with non-missing response
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- DACP Digital: Nelfilcon A digital contact lenses worn bilaterally for 7 days in a daily disposable modality.
- DACP: Nelfilcon A contact lenses worn bilaterally for 7 days in a daily disposable modality.
Arm/Group | DACP Digital | DACP
Number analyzed (Participants) | 60 | 58
logMAR | -0.11 (0.10) | -0.12 (0.09)
Statistical Analysis 1: Comparison: DACP Digital vs DACP; Test type: Non-Inferiority — The pre-specified non-inferiority margin is 0.05. With a sample size of 36 (18 per sequence group), there was approximately 80% power to reject the null hypothesis of inferiority in distance visual acuity with assumed standard deviation of 0.098 for paired difference (one-sided alpha=0.05); Least Squares Mean (LSM) Difference = 0.00, 95% CI 1-sided [upper limit 0.02], Standard Error of Mean 0.008

2. Secondary Outcome: Overall Vision
Description: Subjective rating of overall vision on a scale of 1 (Poor) to 10 (Excellent). Both eyes contributed to the analysis.
Time Frame: Day 7, each product
Population: Full Analysis Set with non-missing response
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DACP Digital | DACP
Number analyzed (Participants) | 59 | 60
units on a scale | 8.8 (1.0) | 8.9 (1.0)
Statistical Analysis 1: Comparison: DACP Digital vs DACP; Test type: Non-Inferiority — The pre-specified non-inferiority margin is 1.0. With a sample size of 48 (24 per sequence group), there was approximately 80% power to reject the null hypothesis of inferiority in subjective overall vision with assumed standard deviation of 2.29 for paired differences (one-sided alpha=0.05); LSM Difference = -0.0, 95% CI 1-sided [lower limit -0.3], Standard Error of Mean 0.15

ADVERSE EVENTS:
Time Frame: Dispense through study completion, an average of 14 days
Description: Adverse Events were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol. This analysis population includes all subjects/eyes that were exposed to any study lenses in the study (Safety Analysis Set), based on treatment-specific exposure.
Groups:
- DACP Digital: All subjects exposed to nelfilcon A digital contact lenses
- DACP: All subjects exposed to nelfilcon A contact lenses
Arm/Group | DACP Digital | DACP
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/05/NCT03567005/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/05/NCT03567005/SAP_001.pdf